CLINICAL TRIAL: NCT00165126
Title: Dosimetric Analysis of Vaginal Cuff Brachytherapy in Endometrial Carcinoma
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Akila Viswanathan, MD, Dana-Farber Cancer Institute
Other Study IDs: 03-315; NCT00207246 (obsolete NCT alias)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Endometrial Carcinoma; Cervix Cancer; Carcinoma of the Uterus
Keywords: dosimetric analysis; vaginal cuff brachytherapy
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Radiation therapy — Given as standard therapy

SUMMARY:
The purpose of this study is to investigate the effect of certain variables such as the fullness of the patients bladder and the position of the treatment applicator on the dose of radiation that other organs such as the bladder and the rectum receive during radiation treatment for endometrial carcinoma.

DETAILED DESCRIPTION:
* This study is separated into 2 phases. In phase 1, patients will be asked to have their bladder full for the second planned insertion of the brachytherapy applicator and empty for the third insertion. For phase 2, the effect of cylinder angle on normal tissue dosimetry will be investigated. Of the two bladder states assessed in phase 1 (empty or full), the one deemed to give the lower dose to the total amount of bladder tissue will be considered the standard and applied to all patients in phase 2.
* In phase 1, to standardize bladder filling, patients will be asked to empty their bladder, then to drink 32 oz of water one and a half hours before the CT scan. The patient will undergo a treatment-planning scan after the brachytherapy cylinder is inserted and before brachytherapy treatment.
* In phase 2, patients will be asked to fill or empty their bladder according to the results of phase 1. The vaginal cylinder will be placed horizontally for the second treatment. The cylinder will then be angled at a specific angle for the subsequent treatment.
* A history and physical exam will be performed within 2 weeks of study entry, then at 14 days, 90 days, and 180 days following the completion of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of carcinoma of the uterus, post-hysterectomy stages I-IVA or vaginal cuff recurrence. Or post-hysterectomy cervix cancer stages IA or IB or post hysterectomy vaginal cancer stage I.
* ECOG performance status of less than or equal to 2
* 18 years of age or older

Exclusion Criteria:

* Distant metastases
* Inoperable disease

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with carcinoma of the uterus, post-hysterectomy stages I-IVA or vaginal cuff recurrence or post-hysterectomy cervix cancer stages IA or IB or post hysterectomy vaginal cancer stage I that will be undergoing radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2004-01; Primary Completion 2006-01 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akila Viswanathan, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute/Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts